CLINICAL TRIAL: NCT00095368
Title: A Phase III, Randomized, Double-Blind, Double-Dummy Multicenter Study to Evaluate the Efficacy and Safety of 775 mg APC-111 MP Tablet QD for 7 Days vs Penicillin VK 250 mg QID for 10 Days in Patients With Streptococcus Pyogenes
Brief Title: APC-111 Once a Day (QD) for 7 Days vs. Penicillin Taken Four Times a Day (QID) for 10 Days in Patients With Strep Throat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advancis Pharmaceutical Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111.301
Record Dates: First submitted 2004-11-03; First posted 2004-11-04 (Estimated); Last update posted 2006-12-08 (Estimated); Status verified 2005-04

CONDITIONS: Pharyngitis; Tonsillitis
Keywords: Pharyngitis; Tonsillitis
MeSH Terms: conditions — Pharyngitis; Tonsillitis | interventions — Pharmaceutical Preparations

INTERVENTIONS:
Drug: Amoxicillin Pulsatile Release Multiparticulate Tablet (drug)

SUMMARY:
The purpose of the this study is to evaluate the safety of efficacy of APC-111 775 mg MP tablet once daily dosing for 7 days for treating patients with strep throat. The evaluation will look to confirm if APC-111 eliminates the bacterial infection (Streptococcus pyogenes).

ELIGIBILITY:
Inclusion Criteria:

* Give informed consent, assent and patient authorization
* Age 12 and over
* A clinical diagnosis of acute pharyngitis or tonsillitis
* A positive rapid Strep test
* Can swallow the oral study dosage forms
* Females must have a negative urine pregnancy test and be using acceptable birth control if sexually active

Exclusion Criteria:

* Chronic or recurrent odynophagia
* Need for hospitalization or IV antimicrobial therapy
* Pharyngitis known or suspected due to a pathogen resistant to beta-lactam antimicrobials
* Known carrier of S. pyogenes
* Allergies to penicillin or other beta-lactam antibiotics
* Any serious illness or concomitant condition that the investigator judges will preclude inclusion to the study
* Seizure disorder
* Pregnant or nursing
* Expectation of additional systemic antibacterials would be required for another condition
* Current drug or alcohol abuse
* Any experimental drug or device within the last 30 days
* Prior systemic antibiotic therapy within the last 30 days
* Hospitalization within the last month which included antibacterial therapy
* The presence of clinically significant hematologic conditions, etc
* Probenecid treatment

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 2004-10; Study Completion 2005-05

PRIMARY OUTCOMES:
Bacteriological outcome at the Test of Cure Visit

SECONDARY OUTCOMES:
Bacteriological outcome at the Late Post Therapy Visit
Clinical Outcome
Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Manford Gooch, MD, Salt Lake City, Utah, United States